CLINICAL TRIAL: NCT04720534
Title: A Double-Blind, Placebo-Controlled Phase 2b Study to Evaluate the Efficacy and Safety of ARO-APOC3 in Adults With Severe Hypertriglyceridemia
Brief Title: Study to Evaluate ARO-APOC3 in Adults With Severe Hypertriglyceridemia
Acronym: SHASTA-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROAPOC3-2001
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Severe Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- ARO-APOC3 10 mg, Day 1 and Week 12 (Experimental): 2 doses of ARO-APOC3 by subcutaneous (sc) injection
  Interventions: Drug: ARO-APOC3
- ARO-APOC3 25 mg, Day 1 and Week 12 (Experimental): 2 doses of ARO-APOC3 by sc injection
  Interventions: Drug: ARO-APOC3
- ARO-APOC3 50 mg, Day 1 and Week 12 (Experimental): 2 doses of ARO-APOC3 by sc injection
  Interventions: Drug: ARO-APOC3
- Placebo, Day 1 and Week 12 (Placebo Comparator): calculated volume to match active treatment by sc injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARO-APOC3 — 2 doses of ARO-APOC3 by subcutaneous (sc) injection
  Arms: ARO-APOC3 10 mg, Day 1 and Week 12; ARO-APOC3 25 mg, Day 1 and Week 12; ARO-APOC3 50 mg, Day 1 and Week 12
Drug: Placebo — calculated volume to match active treatment by sc injection
  Arms: Placebo, Day 1 and Week 12

SUMMARY:
The purpose of AROAPOC3-2001 is to evaluate the efficacy and safety of ARO-APOC3 in participants with severe hypertriglyceridemia. Participants will receive 2 subcutaneous injections of ARO-APOC3.

ELIGIBILITY:
Inclusion Criteria:

* Based on medical history, evidence of TG ≥ 500 mg/dL and ≤ 4000 mg/dL at Screening
* Fasting TG ≥ 500 mg/dL at Screening
* Willing to follow diet counseling per Investigator judgment based on local standard of care
* Women of childbearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be willing to use contraception
* Willing to provide written informed consent and to comply with study requirements

Exclusion Criteria:

* Active pancreatitis within 12 weeks prior to first dose
* Any planned bariatric surgery or similar procedures to induce weight loss from consent to end of study
* Acute coronary syndrome event within 24 weeks of first dose
* Major surgery within 12 weeks of first dose
* Planned coronary intervention (e.g., stent placement or heart bypass) or any non-cardiac major surgical procedure throughout the study
* Uncontrolled hypertension
* Human immunodeficiency virus (HIV) infection, seropositive for Hepatitis B (HBV), seropositive for Hepatitis C (HCV)
* Uncontrolled hypothyroidism or hyperthyroidism
* Hemorrhagic stroke within 24 weeks of first dose
* Malignancy within the last 2 years prior to date of consent requiring systemic treatment (some exceptions apply)

Note: additional inclusion/exclusion criteria may apply per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in Fasting Triglycerides (TG) at Week 24 | Baseline, Week 24

SECONDARY OUTCOMES:
Percent Change from Baseline in Fasting TG Over Time Through Week 48 | Baseline, up to Week 48
Percent Change from Baseline in Apolipoprotein (Apo)C-III at Week 24 | Baseline, Week 24
Percent Change from Baseline in ApoC-III Over Time Through Week 48 | Baseline, up to Week 48
Percent Change from Baseline in Fasting Non-High-Density Lipoprotein-Cholesterol (Non-HDL-C) at Week 24 | Baseline, Week 24
Percent Change from Baseline in Fasting Non-HDL-C Over Time Through Week 48 | Baseline, up to Week 48
Percent Change from Baseline in Fasting High-Density Lipoprotein-Cholesterol (HDL-C) at Week 24 | Baseline, Week 24
Percent Change from Baseline in Fasting HDL-C Over Time Through Week 48 | Baseline, up to Week 48
Percent Change from Baseline in Fasting Total Apolipoprotein B (ApoB) at Week 24 | Baseline, Week 24
Percent Change from Baseline in Fasting Total ApoB Over Time Through Week 48 | Baseline, up to Week 48
Percent Change from Baseline in Fasting Low-density Lipoprotein-Cholesterol (LDL-C) Using Ultracentrifugation | Baseline, Week 24
Percent Change from Baseline in Fasting LDL-C Using Ultracentrifugation Over Time Through Week 48 | Baseline, up to Week 48
Change from Baseline in Plasma Concentration of ARO-APOC3 Over Time Through Week 48 | Baseline, up to Week 48
Number of Participants with Adverse Events (AEs) and/or Serious Adverse Events (SAEs) Possibly or Probably Related to Treatment | up to Week 48

CONTACTS AND LOCATIONS:
Locations (74):
- United States (33):
  - Research Site 2, Beverly Hills, California
  - Research Site 4, Palm Springs, California
  - Research Site 5, Boca Raton, Florida
  - Research Site 6, Fort Lauderdale, Florida
  - Research Site 10, Miami, Florida
  - Research Site 9, Miami, Florida
  - Research Site 11, Miami, Florida
  - Research Site 8, Miami, Florida
  - Research Site 12, Miami Springs, Florida
  - Research Site 14, Port Orange, Florida
  - Research Site 16, Dunwoody, Georgia
  - Research Site 17, Arlington Heights, Illinois
  - Research Site 18, Lexington, Kentucky
  - Research Site 20, Minneapolis, Minnesota
  - Research Site 21, Tupelo, Mississippi
  - Research Site 22, Kalispell, Montana
  - Research Site 23, Omaha, Nebraska
  - Research Site 24, Las Vegas, Nevada
  - Research Site 25, Long Island City, New York
  - Research Site 26, New Windsor, New York
  - Research Site 27, New York, New York
  - Research Site 29, Morehead City, North Carolina
  - Research Site 30, Fargo, North Dakota
  - Research Site 31, Dayton, Ohio
  - Research Site 32, Franklin, Ohio
  - Research Site 33, Maumee, Ohio
  - Research Site 34, Oklahoma City, Oklahoma
  - Research Site 35, Greenville, South Carolina
  - Research Site 36, Chattanooga, Tennessee
  - Research Site 38, Houston, Texas
  - Research Site 39, Houston, Texas
  - Research Site 40, San Antonio, Texas
  - Research Site 41, Manassas, Virginia
- Australia (6):
  - Research Site 43, Perth, Nedlands
  - Research Site 42, Camperdown, New South Wales
  - Research Site 44, Brisbane, Queensland
  - Research Site 45, Sippy Downs, Queensland
  - Research Site 46, Adelaide, South Australia
  - Research Site 47, Clayton, Victoria
- Canada (6):
  - Research Site 49, Concord, Ontario
  - Research Site 50, London, Ontario
  - Research Site 51, Toronto, Ontario
  - Research Site 52, Chicoutimi, Quebec
  - Research Site 53, Greenfield, Quebec
  - Research Site 54, Montreal, Quebec
- Germany (2):
  - Research Site 55, Aachen
  - Research Site 56, Leipzig
- Hungary (9):
  - Research Site 57, Baja
  - Research Site 58, Baja
  - Research Site 59, Balatonföldvár
  - Research Site 60, Békéscsaba
  - Research Site 61, Debrecen
  - Research Site 62, Gyöngyös
  - Research Site 63, Komárom
  - Research Site 65, Nyíregyháza
  - Research Site 64, Nyíregyháza
- Netherlands (3):
  - Research Site 66, Amsterdam
  - Research Site 67, Dordrecht
  - Research Site 68, Sneek
- New Zealand (5):
  - Research Site 73, Grafton, Auckland
  - Research Site 69, Christchurch
  - Research Site 70, Hamilton
  - Research Site 71, Papatoetoe
  - Research Site 72, Rotorua
- Poland (10):
  - Research Site 74, Bydgoszcz
  - Research Site 75, Elblag
  - Research Site 76, Gdynia
  - Research Site 83, Lodz
  - Research Site 78, Oświęcim
  - Research Site 79, Poznan
  - Research Site 80, Puławy
  - Research Site 81, Rzeszów
  - Research Site 82, Wołomin
  - Research Site 77, Łęczyca

REFERENCES:
- [Derived] Gaudet D, Pall D, Watts GF, Nicholls SJ, Rosenson RS, Modesto K, San Martin J, Hellawell J, Ballantyne CM. Plozasiran (ARO-APOC3) for Severe Hypertriglyceridemia: The SHASTA-2 Randomized Clinical Trial. JAMA Cardiol. 2024 Jul 1;9(7):620-630. doi: 10.1001/jamacardio.2024.0959. PMID 38583092